CLINICAL TRIAL: NCT03045562
Title: Effects of Salvianolate Injection on Myocardial Microcirculation in Patients With Acute ST Segment Elevation Myocardial Infarction After Primary PCI
Brief Title: Effects of Salvianolate Injection on Myocardial Microcirculation in Patients With Acute STEMI After Primary PCI
Acronym: SISTEMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Valley Group of China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GV-MD-CT201602
Record Dates: First submitted 2017-01-20; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Saline Solution; Sodium Chloride; salvianolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Patients will be assigned to receive 100ml of normal saline
  Interventions: Drug: Normal saline
- Experimental group (Experimental): Patients will be assigned to receive Salvianolate injection dissolved in 100ml of normal saline
  Interventions: Drug: Salvianolate injection

INTERVENTIONS:
Drug: Normal saline — Patients will be assigned to receive 100ml of normal saline in catherter room setting,and following similar medicine once daily for 7 days.
  Other Names: 0.9% sodium chloride solution
  Arms: Control group
Drug: Salvianolate injection — Patients will be assigned to receive Salvianolate injection dissolved in 100ml of normal saline in catherter room setting,and following similar medicine once daily for 7 days.
  Other Names: Salvianolate
  Arms: Experimental group

SUMMARY:
To evaluate the influence of Salvianolate injection on myocardial microcirculation perfusion in subjects with STEMI who underwent primary PCI

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind and controlled study.536 subjects of STEMI who underwent primary PCI within the first 12 hours will be enrolled.all patients were assigned to receive 300mg of asprin and ≥300mg of clopidogrel as loading dose,and following 100mg and 75mg once daily respectively.Patients were assigned to receive Salvianolate injection or 0.9% sodium chloride injection in catherter room setting,and following similar medicine once daily respectively for 7 days.Myocardial circulation perfusion will be checked with mmediate coronary angiography parameters,ECG,echocardiographic，CK-MB.The major adverse cardiovascular events will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent must be obtained prior to any study procedure.
2. Age>18 years.
3. Subjects of STEMI who underwent primary PCI within the first 12 hours.

Exclusion Criteria:

1. Allergic to Salvianolate injection
2. Mechanical complications
3. History of severe renal or hepatic insufficiency
4. Pregnant or breastfeeding women
5. Pool compliance,greater risks result from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
TIMI flow grade | an average of 2 hours
  Use TIMI flow grade to evaluate myocardial circulation perfusion
TIMI myocardial perfusion grade | an average of 2 hours
  Use TIMI myocardial perfusion grade to evaluate myocardial circulation perfusion

SECONDARY OUTCOMES:
ST-segment resolution | up to 90 minutes
  Use ST-segment resolution to evaluate the epicardial blood flow perfusion
myocardial contrast echocardiograph | up to 7 days
  Use myocardial contrast echocardiograph to evaluate the myocardial microcirculation perfusion
creatine kinase isoenzyme | up to 48 hours
  Use creatine kinase isoenzyme to evaluate myocardial infarct size
major adverse cardiovascular events | an average of 30 days
  all-caused death, re-infarction, target vessel revascularization, stroke

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, doctor, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China